CLINICAL TRIAL: NCT01690689
Title: Investigation of a Customized Femoral Resurfacing Implant (Episealer® Knee Condyle Device) to Assess the Safety Profile and Performance for 2 Years Post-operatively
Brief Title: Investigation of a Customized Femoral Resurfacing Implant
Acronym: Knee100
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Episurf Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCR-120412-01
Record Dates: First submitted 2012-08-10; First posted 2012-09-24 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Articular Cartilage Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery (Experimental): Implant surgery
  Interventions: Device: Implant surgery

INTERVENTIONS:
Device: Implant surgery — surgery

SUMMARY:
The purpose is to assess the safety profile and performance of a femoral resurfacing implant for localized chondral lesions.

DETAILED DESCRIPTION:
The implant's safety profile will be assessed by incidence of any subject having any of the seven identified implant-related clinical undesirable side effects. This will be analyzed with a one-side exact binomial test on significance level 0.05, at 24 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 30 ≤ 65 years
3. Chondral defects of the femoral cartilage ICRS grade 3 (severely abnormal cartilage defects > 50% of the cartilage depth) or grade 4 (severely abnormal, through the cartilage depth) on medial or lateral femoral condyles
4. Cartilage lesion area < 3.2 cm2 (diameter < 2 cm)
5. Failed earlier conservative or surgical interventions such as lavage, abrasions, drilling or microfracture
6. VAS-pain symptom >40 for more than 6 months
7. The arthroscopic finding corresponds to the expected; size of cartilage lesion is correct and no other significant pathology (see CIP, "Intra-operative check-list", Appendix I)
8. Capable of completing self-administered questionnaires
9. Willing to comply with the follow-up requirements of the study
10. Signed informed consent

Exclusion Criteria:

1. BMI ≥ 35 kg/m2 (severe obesity)
2. Instability or deficiency of soft tissues, vascular or muscular insufficiency
3. Metabolic disorders which may impair bone formation
4. Diabetes mellitus
5. Smokers
6. Diagnosis of a concomitant knee injury which the Investigator appreciates may interfere with study participation (i.e. may confound efficacy assessment or healing at the involved knee joint level)
7. Irresolvable joint pain or loss-of-function with an undeterminable cause
8. Diagnosis of a concomitant meniscal injury in involved knee that requires surgical intervention
9. Loss of joint space on standing radiographs (≥ 1 on Ahlbäck-scale (0-5))
10. Avascular necrosis
11. Infections, systemic or local
12. Known metal allergies
13. History of inflammatory arthritis
14. Pregnancy
15. Pacemaker implant
16. History of drug or substance abuse
17. Systemic administration within 30 days prior to the study of any type of corticosteroid, antineoplastics, immune stimulating or immunosuppressive agents
18. Participation in another clinical trial using an investigational new drug or device within 30 days of entrance into this study.
19. Condition that may have an impact on the outcome of the investigation as judged by the Investigator.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 24 months
  The primary efficacy analysis in this study is to ascertain that the incidence of at least one subject having any of the seven identified clinical undesirable side effects is lower than 38 % (risk profile of the comparator) up to the 24 months analysis in the PP population. This will be analyzed with a one-side exact binomial test on significance level 0.05

SECONDARY OUTCOMES:
Clinical performance | 24 months
  Clinical performance, by questionnaires and knee ROM measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Zetterberg, Study Director — Episurf Medical
Locations (3):
- Sweden (3):
  - Lund University Hospital, Department of Ortopedics, Lund
  - Aleris Specialistvård, Stockholm
  - Sports Medicine Umeå, Umeå